CLINICAL TRIAL: NCT05761288
Title: Microbreaks and Intraoperative Exercises for Gynecologic Surgeons (MIGS Trial)
Brief Title: Intraoperative Exercises & Musculoskeletal Pain in Gynecologic Surgeons
Acronym: GynIEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 00002946
Record Dates: First submitted 2023-02-08; First posted 2023-03-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Work-related Injury; Physical Injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Once participants are enrolled, all participant surgery days will be assessed for inclusion based on the inclusion criteria above. Surgery days will be randomized to surgery days with microbreaks and exercises and surgery days without microbreaks and exercises. The surgeon will be informed of the randomization assignment prior to the surgery day.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery days with intraoperative microbreaks and exercises (Experimental): Surgery days randomized to intraoperative microbreaks and exercises will include standardized breaks lasting approximately 1.5-2 minutes. During these breaks, surgeons will perform a set of targeted stretches or exercises while remaining sterile. The exercises will be performed just before surgical time-out, at a surgically safe and convenient time 45-75 mins after the start of the case and at the end of the case. A surgically safe and convenient time means the surgeon feels that it is safe to take an approximately 1.5-2 minute break during the procedure at that time. Surgeons will skip the microbreak if there is no surgically convenient or safe time during the case. Surgeons will stop the microbreak at any point if needed to ensure patient safety.
  Interventions: Behavioral: Intraoperative microbreaks and exercises
- Surgery days without intraoperative microbreaks and exercises (No Intervention): Surgery days without intraoperative microbreaks and exercises will include no intervention. Surgeons will perform the surgeries as they are normally performed and surgeons will not take microbreaks or perform exercises.

INTERVENTIONS:
Behavioral: Intraoperative microbreaks and exercises — Intraoperative microbreaks and exercises will include standardized breaks lasting approximately 1.5-2 minutes. During these breaks, surgeons will perform a set of targeted stretches or exercises while remaining sterile. Intervention exercises include: chest and shoulder opener "elbows in pockets," chin tuck, neck rotation, squat with truncal rotation (chair pose with prayer), and forward bend.
  Arms: Surgery days with intraoperative microbreaks and exercises

SUMMARY:
The goal of this study is to evaluate the effect of intraoperative microbreaks and exercises on gynecologic surgeon body discomfort by conducting a randomized trial. We hypothesize that gynecologic surgeons will experience decreased pain on surgery days with intraoperative microbreaks and exercises without compromising overall surgical performance.

DETAILED DESCRIPTION:
Potential participants include residents, fellows, and attendings performing gynecologic surgery (including benign gynecologists, gynecologic oncologists, minimally invasive gynecologists, and urogynecologists). We will recruit surgeons from the Department of Women's Health at the University of Texas at Austin Dell Medical School. Surgeons will need to have operated on average at least 2 days per month over the last 12 months. Written informed consent will be obtained. Eligible surgery days must include at least one surgery with total operative time of at least 2 hours. Surgeons will be excluded if they are unable to perform the exercises.

Upon agreement to participate in the study, surgeons will complete baseline questionnaires adapted from the standardized Nordic Musculoskeletal Questionnaire (NMSQ) and a survey developed by Plerhoples et al. The NMSQ is a validated questionnaire for the analysis of musculoskeletal symptoms and assesses for history of trouble (ache, pain, discomfort) in body part regions. The survey includes information such as surgeon age, gender, weight, height, dominant hand, surgical volume, years practicing surgery, and activity level.

Once participants are enrolled, all participant surgery days will be assessed for inclusion based on the inclusion criteria above. Surgery days will be randomized to surgery days with microbreaks and exercises and surgery days without microbreaks and exercises. The surgeon will be informed of the randomization assignment prior to the surgery day.

Surgery days randomized to intraoperative microbreaks and exercises will include standardized breaks lasting approximately 1.5-2 minutes. During these breaks, surgeons will perform a set of targeted stretches or exercises while remaining sterile. These exercises were developed with the assistance of a physician specialized in Physical Medicine and Rehab. The exercises will be performed just before surgical time-out, at a surgically safe and convenient time 45-75 mins after the start of the case and at the end of the case. A surgically safe and convenient time means the surgeon feels that it is safe to take an approximately 1.5-2 minute break during the procedure at that time. Surgeons will skip the microbreak if there is no surgically convenient or safe time during the case. Surgeons will stop the microbreak at any point if needed to ensure patient safety. The microbreaks performed during the surgery may add time to the surgery in approximately 1.5-2 minute increments, however prior studies have shown no difference in operative time with addition of microbreaks. Attached is a document outlining the exercises including photos with exercise cues and a video demonstrating the exercises. Participants will have access to these documents before and during the study.

On each surgery day, participating surgeons will complete the "Surgery Day Questionnaire" which will include the Body Part Discomfort (BPD) scale and Surgery Task Load Index (SURG-TLX). The Corlett and Bishop BPD Scale was originally created in 1976 and is a validated technique to assess work-related discomfort by body part regions. Another measure of work-related stress during surgery is the SURG-TLX. This is a validated tool based off the NASA-TLX used to assess overall workload including mental demands, physical demands, temporal demands, task complexity, situational stress, and distractions. At the beginning of all surgery days, the participating surgeon will complete a baseline BPD scale as the first part of the "Surgery Day Questionnaire". Following each surgery day, the surgeon will complete both the BPD scale and the SURG-TLX survey to complete the "Surgery Day Questionnaire" for that day. Participating surgeons are asked to inform the research team if they develop any new work-related injury during the study period.

Data will be collected from medical records about each surgery in the study. The following perioperative data will be collected: surgeries performed, operative time, and intraoperative complications.

At the conclusion of the study, an anonymous exit survey will be performed to give all participants an opportunity to provide feedback. Data will be collected on the results of the exit survey. All data will be collected and stored in our institution's REDcap, a secure electronic application for research.

ELIGIBILITY:
Inclusion Criteria:

* Residents, fellows, and attendings performing gynecologic surgery (including benign gynecologists, gynecologic oncologists, minimally invasive gynecologists, and urogynecologists) who are able to perform the exercises.
* Surgery days must contain at least one gynecologic surgery with two hours of total operating time in one day.
* Surgeons will need to have operated on average at least 2 days per month over the last 12 months.

Exclusion Criteria:

* Participants will be excluded if they are unable to perform the exercises.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Body Part Discomfort (BPD) | On the day of surgery
  On each of the eligible surgery days, we will collect data on body part discomfort and surgical experience using the Body Part Discomfort (BPD) scale. The BPD scale measures body part discomfort using a 10-point scale (1 corresponds with no discomfort and 10 corresponds to maximum body discomfort) for body part regions.

SECONDARY OUTCOMES:
Surgery Task Load Index (SURG-TLX) | On the day of surgery
  The modified SURG-TLX will be evaluated at the end of each surgery day to assess participant experience throughout the surgery day. The SURG-TLX measures 6 areas: mental demands, physical demands, task complexity, situational stress, and distractions.
Perioperative data | On the day of surgery
  surgeries performed, operative time, and intraoperative complications (i.e. bladder/bowel injury, large vessel injury, transfusion, allergic reaction, difficulty ventilating, ICU admission)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corlett EN, Bishop RP. A technique for assessing postural discomfort. Ergonomics. 1976 Mar;19(2):175-82. doi: 10.1080/00140137608931530. No abstract available. PMID 1278144
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Wilson MR, Poolton JM, Malhotra N, Ngo K, Bright E, Masters RS. Development and validation of a surgical workload measure: the surgery task load index (SURG-TLX). World J Surg. 2011 Sep;35(9):1961-9. doi: 10.1007/s00268-011-1141-4. PMID 21597890

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT05761288/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05761288/ICF_001.pdf